CLINICAL TRIAL: NCT00684047
Title: A Prospective, Single-blind, Randomized, Phase II/III Study to Evaluate the Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) as an Adjunct to Hemostasis During Peripheral Vascular Surgery
Brief Title: Safety and Efficacy Study of Fibrin Sealant Grifols Evaluated as an Adjunct to Hemostasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IG402
Record Dates: First submitted 2008-05-20; First posted 2008-05-26 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Target Bleeding Site During Peripheral Vascular Surgery
Keywords: Fibrin Sealant; Hemostasis; Peripheral Vascular Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- FS Grifols Preliminary Part (I) (Experimental): Open label administration of FS Grifols to all subjects
  Interventions: Biological: FS Grifols
- FS Grifols Primary Part (II) (Experimental): Single-blind, randomized (2:1)
  Interventions: Biological: FS Grifols
- Manual Compression Primary Part (II) (Active Comparator): Single-blind, randomized (2:1)
  Interventions: Procedure: Manual Compression

INTERVENTIONS:
Biological: FS Grifols — Fibrin Sealant Grifols (FS Grifols). Preliminary Part (I)
  Arms: FS Grifols Preliminary Part (I)
Biological: FS Grifols — Fibrin Sealant Grifols (FS Grifols). Primary Part (II)
  Arms: FS Grifols Primary Part (II)
Procedure: Manual Compression — Manual Compression. Primary Part (II)
  Arms: Manual Compression Primary Part (II)

SUMMARY:
The purpose of this study is to evaluate the safety and hemostasis effectiveness of human plasma-derived fibrin sealant Grifols (FS Grifols) in peripheral vascular surgery.

DETAILED DESCRIPTION:
The trial consisted of 2 parts: a Preliminary Part (I) and a Primary Part (II). All subjects enrolled in Preliminary Part (I) were treated with FS Grifols. Subjects in Primary Part (II) were randomly allocated in a 2:1 ratio to treatment with FS Grifols or manual compression. The objectives of the study were to evaluate the hemostasis effectiveness of FS Grifols in peripheral vascular surgery and to assess clinical safety, viral safety, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female
* Must be at least 3 years of age with no upper age limit (must be at least 18 years of age in Spain and United Kingdom)
* Require an elective (non-emergency), open (non-laparoscopic; non-endovascular) peripheral vascular surgical procedure
* Have hemoglobin ≥ 9.0 g/dL
* Have platelet count > 70 x 10^3/mm^3
* Required one peripheral vascular procedure involving either an arterial patch angioplasty or an arterial anastomosis utilizing polytetrafluoroethylene or Dacron grafts, according to the Investigator's (the surgeon's) selection:

  1. Carotid endarterectomy requiring patch angioplasty
  2. Carotid-subclavian bypass grafting
  3. Axillo-femoral bypass grafting
  4. Abdominal aortic aneurysm resection and graft replacement
  5. Aorto-mesenteric bypass grafting
  6. Aorto-celiac bypass grafting
  7. Aorto-uni-iliac bypass grafting
  8. Aorto-bi-iliac bypass grafting
  9. Aorto-uni-femoral bypass grafting
  10. Aorto-bi-femoral bypass grafting
  11. Iliac aneurysm resection and graft replacement
  12. Femoral aneurysm resection and graft replacement
  13. Femoral-femoral bypass grafting
  14. Femoral-popliteal bypass grafting
  15. Renal arterial revascularization (bypass grafting)
  16. Renal arterial revascularization (endarterectomy with patch angioplasty)
  17. Popliteal artery revascularization (bypass grafting)
  18. Popliteal artery revascularization (endarterectomy with patch angioplasty)
  19. Femoral endarterectomy with patch angioplasty
  20. Ilio-femoral bypass grafting
* Intra-operative inclusion criterion:

  * A Target bleeding site (TBS)can be identified according to the Investigator's judgment, and the TBS has a mild or moderate arterial bleeding according to the Investigator's judgment

Exclusion Criteria:

* Weighed < 20 kg
* Have a pre-operative (at Baseline Assessments) international normalized ratio ≥ 2.0
* Have a pre-operative (at Baseline Assessments) activated partial thromboplastin time ratio ≥ 1.5
* Have a pre-operative (at Baseline Assessments) serum creatinine > 2 times the upper limit of the normal range
* Were undergoing a re-operative procedure on same arterial patch angioplasty or arterial anastomosis
* Have an infection in the anatomical surgical area
* Have a history of severe (e.g., anaphylactic) reactions to blood or any blood derived product
* Unwilling to receive blood products
* Have positive bleeding history
* Female who was pregnant or nursing
* Are known to abuse alcohol, opiates, psychotropic agents or other chemicals or drugs, or have done so within 12 months to the screening visit.
* Are currently participating in another investigational drug or device clinical study, or have participated within 3 months to the screening visit.
* Were previously included in this clinical trial (protocol number IG402)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-02; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Kozloff, MD, Study Director — Independent
Locations (19):
- Canada (5):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Schulich School of Medicine, London Health Sciences Center, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Spain (6):
  - Hospital Universitario de Getafe, Getafe, Madrid
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de Sabadell, Barcelona
  - Hospital Son Espases, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Edgbaston, Birmingham
  - Frimley Park Hospital, Frimley, Surrey
  - Doncaster Royal Infirmary Hospital, Doncaster
  - Royal Infirmary of Edinburgh, Edinburgh
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - Freeman Hospital, Newcastle upon Tyne
  - St. George's Hospital, Tooting

REFERENCES:
- [Derived] Ma GW, Kucey A, Tyagi SC, Papia G, Kucey DS, Varcoe RL, Forbes T, Neville R, Dueck AD, Kayssi A. The role of sealants for achieving anastomotic hemostasis in vascular surgery. Cochrane Database Syst Rev. 2024 May 2;5(5):CD013421. doi: 10.1002/14651858.CD013421.pub2. PMID 38695613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 20 October 2008 Study Completion Date: 05 May 2014
Groups:
- FS Grifols Preliminary Part (I): FS Grifols was applied in all subjects in this arm. FS Grifols: Fibrin Sealant Grifols (FS Grifols).
- FS Grifols Primary Part (II): FS Grifol was applied in subjects in this arm. FS Grifols: Fibrin Sealant Grifols (FS Grifols).
- Manual Compression Primary Part (II): Manual Compression was applied in subjects in this arm.
Period: Overall Study
Arm/Group | FS Grifols Preliminary Part (I) | FS Grifols Primary Part (II) | Manual Compression Primary Part (II)
Started | 72 | 110 | 57
Completed | 59 | 94 | 52
Not Completed | 13 | 16 | 5

BASELINE CHARACTERISTICS:
Population: Demographic information is summarized for the subjects in the Intent to treat population.
Groups:
- FS Grifols Preliminary Part (I): Subjects treated during FS Grifols Preliminary Part (I) were analyzed. FS Grifols: Fibrin Sealant Grifols (FS Grifols).
- FS Grifols Primary Part (II): Subjects treated during FS Grifols Primary Part (II) were analyzed. FS Grifols: Fibrin Sealant Grifols (FS Grifols).
- Manual Compression Primary Part (II): Subjects treated with manual compression were analyzed.
- Total: Total of all reporting groups
Arm/Group | FS Grifols Preliminary Part (I) | FS Grifols Primary Part (II) | Manual Compression Primary Part (II) | Total
Number analyzed (Participants) | 72 | 110 | 57 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.91) | 68.4 (8.90) | 67.0 (10.28) | 68.0 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 18 | 50
  Male | 55 | 95 | 39 | 189

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is Time to Hemostasis.
Description: The primary efficacy endpoint of the study is time to hemostasis (TTH), measured in minutes from the start of treatment application (TStart) at the TBS to the achievement of hemostasis at that site or to the end of the 10-minute observational period if hemostasis has not yet been achieved.
Time Frame: The start of treatment application at the target bleeding site (TBS) to the achievement of hemostasis at that site or to the end of the 10-minute observational period when the hemostasis has not yet been achieved.
Measure: Number; unit: percentage of subjects
Groups:
- FS Grifols Primary Part (II): FS Grifols was applied during FS Grifols Primary Part (II). FS Grifols: Fibrin Sealant Grifols (FS Grifols).
- Manual Compression Primary Part (II): Manual compression was applied during the Manual Compression Primary Part (II).
Arm/Group | FS Grifols Primary Part (II) | Manual Compression Primary Part (II)
Number analyzed (Participants) | 110 | 57
percentage of subjects
  TTH ≤ 3 minutes (cumulative, % ) | 46.4 | 26.3
  TTH ≤ 4 minutes (cumulative, %) | 62.7 | 31.6
  TTH ≤ 5 minutes (cumulative, %) | 74.5 | 49.1
  TTH ≤ 7 minutes (cumulative, %) | 79.1 | 56.1
  TTH ≤ 10 minutes (cumulative, %) | 88.2 | 71.9
  Treatment Failure | 11.8 | 28.1

2. Secondary Outcome: Proportions of Subjects Achieving Hemostasis
Description: The cumulative proportions of subjects who achieved hemostasis during the 10- minute observation period in Primary Part (II)
Time Frame: 10 minutes from the start of treatment application at the target bleeding site
Population: intent to treat population
Measure: Number; unit: percentage of participants
Groups:
- FS Grifols Primary Part (II): FS Grifol was applied in subjects. FS Grifols: Fibrin Sealant Grifols (FS Grifols).
Arm/Group | FS Grifols Primary Part (II) | Manual Compression Primary Part (II)
Number analyzed (Participants) | 110 | 57
percentage of participants | 88.2 | 71.9

3. Secondary Outcome: Prevalence of Treatment Failures
Description: The cumulative proportions of subjects who did not achieve hemostasis during the 10- minute observation period in Primary Part (II)
Time Frame: 10 minutes from the start of treatment application at the target bleeding site
Population: intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | FS Grifols Primary Part (II) | Manual Compression Primary Part (II)
Number analyzed (Participants) | 110 | 57
percentage of participants | 11.8 | 28.1

ADVERSE EVENTS:
Time Frame: Six weeks
Groups:
- FS Grifols [Pooled Preliminary Part (I) + Primary Part (II)]: The safety population included all subjects treated with FS Grifols in Preliminary Part (I) and Primary Part (II). FS Grifols: Fibrin Sealant Grifols (FS Grifols): Preliminary Part (I): 72 subjects and Primary Part (II): 110 subjects.
  The safety population included five additional subjects treated with FS Grifols instead of manual compression who were not included in the baseline and efficacy outcome analyses.
- Manual Compression Primary Part (II): The safety population included all subjects treated with manual compression in the Manual Compression Primary Part (II). Five subjects randomized to this arm were treated with FS Grifols and thus were removed from this arm for the safety analyses.
Arm/Group | FS Grifols [Pooled Preliminary Part (I) + Primary Part (II)] | Manual Compression Primary Part (II)
Serious Adverse Events (participants affected / at risk) | 47/187 | 9/52
Other Adverse Events (participants affected / at risk) | 151/187 | 45/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS Grifols [Pooled Preliminary Part (I) + Primary Part (II)] (N=187) | Manual Compression Primary Part (II) (N=52)
Post Operative Wound Infection (Infections and infestations) | 4 (4) | 1 (1)
Wound Infection (Infections and infestations) | 3 (3) | 2 (2)
Abdominal Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardio-respiratory Arrest (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Chronic (Cardiac disorders) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Operative Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Graft Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 2 (3) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 2 (2) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial Eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Multiorgan Failure (General disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FS Grifols [Pooled Preliminary Part (I) + Primary Part (II)] (N=187) | Manual Compression Primary Part (II) (N=52)
Procedural Pain (Injury, poisoning and procedural complications) | 112 (113) | 36 (36)
Nausea (Gastrointestinal disorders) | 44 (51) | 10 (11)
Constipation (Gastrointestinal disorders) | 39 (39) | 8 (8)
Vomiting (Gastrointestinal disorders) | 14 (25) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 13 (13) | 3 (3)
Hypotension (Vascular disorders) | 32 (34) | 8 (8)
Blood Potassium Decreased (Investigations) | 12 (13) | 5 (5)
Pyrexia (General disorders) | 14 (15) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 11 (12) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 8 (8) | 3 (4)
Hypertension (Vascular disorders) | 7 (7) | 3 (3)
Haematoma (Vascular disorders) | 7 (8) | 3 (4)
Blood Magnesium Decreased (Investigations) | 5 (5) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 3 (3)
Oedema Peripheral (General disorders) | 9 (9) | 5 (5)
Insomnia (Psychiatric disorders) | 7 (7) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 16 (17) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor at least thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsor's request, Site will remove any Confidential Information (other than Study results), and incorporate all reasonable comments by Sponsor, or delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor's Inventions.